CLINICAL TRIAL: NCT01445392
Title: A Phase 1, Single Center, Dose-Escalation Study of SS1(dsFv)PE38 Administered Concurrently With Pemetrexed and Cisplatin in Subjects With Unresectable Malignant Epithelial Pleural Mesothelioma
Brief Title: SS1(dsFV)PE38 Plus Pemetrexed and Cisplatin to Treat Malignant Pleural Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080026; 08-C-0026; NCT00575770 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08-01

CONDITIONS: Mesothelioma
Keywords: Recombinant Immunotoxin; Monoclonal Antibody; Pseudomonas Exotoxin; Targeted Therapy; Pleural Mesothelioma; Mesothelioma; Epithelial Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- 1 (Experimental): Multi-cycle cohort
  Interventions: Biological: Multicycle SS1P; Drug: Pemetrexed; Drug: Cisplatin
- 2 (Experimental): Single cycle cohort
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Biological: Single cycle SS1P

INTERVENTIONS:
Biological: Multicycle SS1P — Assigned dose level of SS1(dsFv)PE38 on days 1, 3 & 5 of a 21 day cycle for 2 cycles
  Arms: 1
Drug: Pemetrexed — 500 mg/m^2 on day 1 of each 21 day cycle until disease progression
Drug: Cisplatin — 75 mg/m^2 on day 1 of each 21 day cycle until disease progression
Biological: Single cycle SS1P — Patients 1 - 3 of single cycle cohort. 45 mcg/kg of SS1(dsFv)PE38 on 4 or 5 days (depending on dose level) of cycle 1 only.
  Arms: 2

SUMMARY:
Background:

Standard therapy for mesothelioma is a combination of the drugs pemetrexed and cisplatin. However, the benefits of this treatment are limited, and in most treated patients the disease continues to worsen.

SS1(dsFV)PE38 is a genetically engineered drug. It contains an antibody that binds to a certain protein on mesothelioma cells and a toxin (type of poison) made from a product of a bacterium called Pseudomonas aeruginosa. It is hoped that the antibody will attach to the cancer cells, allowing the toxin to enter and kill the cells.

Objectives:

To find out if SS1(dsFV)PE38, together with pemetrexed and cisplatin is safe and tolerable in patients with mesothelioma.

To determine the maximum tolerated dose of SS1(dsFV)PE38 (the highest dose that does not cause unacceptable side effects).

To see if SS1(dsFV)PE38 given with pemetrexed and cisplatin has any effect on patients tumors.

To learn how the body breaks down SS1(dsFV)PE38.

Eligibility:

Patients 18 years of age and older with epithelial pleural mesothelioma whose disease cannot be cured with surgery, and have not had prior treatment with chemotherapy.

Design:

Treatment with pemetrexed, cisplatin and SS1(dsFV)PE38 in two 21-day cycles as follows:

* Day 1 - Intravenous (through a vein) infusions of pemetrexed and cisplatin.
* Days 1 and 2 - Intravenous solution to prevent dehydration that might occur with SS1(dsFV)PE38.
* Days 1, 3 and 5 Intravenous infusion of SS1(dsFV)PE38. Small groups (3 to 6) of patients are given SS1(dsFV)PE38 at a certain dose level. If the first group experiences no significant side effects, the next group a higher dose. This continues in succeeding groups until the maximum tolerated study dose (highest dose that patients can be given safely) is determined.

Continuing standard treatment with additional cycles of pemetrexed and cisplatin.

Evaluations during the treatment period:

* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Questions about medications and side effects.
* Blood and urine tests.
* Disease evaluation with CT, chest X-ray, and possibly PET scans, lung function tests, pulse oximetry, performance of daily activities and quality-of-life questionnaires.

Post-treatment evaluations:

* Clinic visits at months 1, 3, 6, 12, 15, 18 and 21 for physical examination and disease assessment.
* End-of-study visit for blood tests, vital signs and weight measurements, disease assessment, electrocardiogram, pregnancy test for women who can become pregnant

DETAILED DESCRIPTION:
Background:

SS1P (dsFv) PE38, is a recombinant immunotoxin targeting the tumor antigen mesothelin that is highly expressed in malignant mesothelioma. The maximum tolerated dose (MTD) of SS1 dsFv has been established in a phase I study.

Combination therapy with pemetrexed plus cisplatin is the standard first line therapy for malignant mesothelioma, but results in a median overall survival of only 12.1 months.

Combination of SS1(dsFv)PE38 with pemetrexed plus cisplatin could result in improved outcomes for patients with mesothelioma.

Objectives:

To determine the MTD of SS1(dsFv)PE38 that can be safely administered in combination with pemetrexed plus cisplatin in patients with mesothelioma.

To characterize the toxicity profile of SS1(dsFv)PE38.

To study the pharmacokinetics of SS1(dsFv)PE388.

To observe anti-tumor activity, if any of SS1(dsFv)PE38 in combination with pemetrexed plus cisplatin.

Eligibility:

Subjects with histologically confirmed epithelial pleural mesothelioma.

No prior radiotherapy (except palliative localized radiotherapy),systemic chemotherapy or biologic therapy for pleural mesothelioma.

Design:

This is a phase I dose-escalation study of SS1(dsFv)PE38 in combination with pemetrexed plus cisplatin.

The dose of pemetrexed plus cisplatin will be the standard dose approved for malignant mesothelioma. The dose of SS1(dsFv)PE38 will be escalated to find the safe dose in combination with pemetrexed plus cisplatin.

SS1(dsFv)PE38 will be administered concurrently with pemetrexed plus cisplatin in cycles one and two, and subjects will receive additional cycles of pemetrexed and cisplatin as per standard practice.

Patients will be assessed for response every 6 weeks.

An additional Single Cycle of SS1(dsFv)PE38 Cohort will involve up to 16 patients who will receive SS1(dsFv)PE38 administered for four or five doses during the first cycle concurrently with pemetrexed and cisplatin; subjects in this cohort will receive additional

cycles of pemetrexed and cisplatin as per standard practice

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must meet all of the following criteria to be eligible to participate in the study:

Subjects must have histologically confirmed epithelial or biphasic pleural mesothelioma not amenable to potentially curative surgical resection. However, patients with biphasic tumors that have a predominantly sarcomatoid component will be excluded.

Measurable disease

Subjects must be greater than or equal to 18 years old

Karnofsky Performance Status (KPS) of greater than or equal to 70

Life expectancy of greater than 3 months, as assessed by the principal investigator.

Adequate organ function with:Hepatic function: serum transaminases (either ALT or AST) or bilirubin, less than or equal to Grade 1, unless due to cancer or Gilbert s disease; less than or equal to Grade 2, if due to cancer

Renal function: serum creatinine clearance greater than or equal to 60mL/min as estimated by Cockroft-Gault formula.

Bone marrow function: ANC of at least 1,500/mm (3), Platelet count at least 100,000/mm (3)

Pulmonary Function: FEV (1) greater than or equal to 50 percent of predicted value (post-pleural drainage and bronchodilation if these are indicated)

Must be able to understand and sign informed consent

Female and male subjects agree to use an approved method of contraception during the study

EXCLUSION CRITERIA:

Subjects must not be pregnant or breast feeding

Prior radiotherapy (except palliative extra-thoracic localized radiotherapy) or biologic therapy for malignant pleural mesothelioma within 4 weeks

Prior systemic chemotherapy for malignant pleural mesothelioma

Documented and ongoing central nervous system involvement with their malignant disease (history of CNS involvement is not an exclusion criterion but the CNS metastases should have been adequately treated (radiation or surgical resection) and subjects are free from symptoms for 3 months off steroids).

Clinically significant heart disease (New York Heart Association Class III or IV)

Active bacterial or fungal infection.

Baseline coagulopathy greater than or equal to Grade 3 unless due to anticoagulant therapy

Surgery or pleurodesis within 2 weeks

HIV positive serology (due to increased risk of severe infection and unknown interaction of SS1(dsFv)PE38 with antiretroviral drugs)

Hepatitis B surface antigen positivity

Subjects with other (non-mesothelioma) cancers who meet eligibility criteria and have had less than 5 years of disease-free survival will be considered on a case-by-case basis

Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11-14; Primary Completion 2014-01-31 (Actual); Study Completion 2016-10-03 (Actual)

PRIMARY OUTCOMES:
Safety and MTD | 30 days after last dose
  list of adverse events and highest dose at which fewer than 2 subjects experienced DLT
Best overall response | Assessed every 42 days until disease progression
  proportion of subjects experiencing complete response, partial response or stable disease as a best overall response

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chang K, Pastan I. Molecular cloning of mesothelin, a differentiation antigen present on mesothelium, mesotheliomas, and ovarian cancers. Proc Natl Acad Sci U S A. 1996 Jan 9;93(1):136-40. doi: 10.1073/pnas.93.1.136. PMID 8552591
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Hassan R, Kreitman RJ, Pastan I, Willingham MC. Localization of mesothelin in epithelial ovarian cancer. Appl Immunohistochem Mol Morphol. 2005 Sep;13(3):243-7. doi: 10.1097/01.pai.00000141545.36485.d6. PMID 16082249